CLINICAL TRIAL: NCT03602703
Title: Detection of Immune Cell Responses in Chronic HCV Patients Developing Hepatocellular Carcinoma After Treatment With Direct Acting Antiviral Drugs (DAAs)
Brief Title: Immune Responses in Hepatocellular Carcinoma Patients After Treatment With Direct Acting Antiviral Drugs
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidi Karam, Lecturer, Assiut University
Other Study IDs: 17300211
Record Dates: First submitted 2018-07-03; First posted 2018-07-27 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2018-07

CONDITIONS: Drug-Induced Liver Injury
Keywords: Direct acting antiviral drugs immune responses
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) will be isolated using ficoll gradient method and will then be stored at -80C. Plasma will be isolated and stored at - 20C and further analysis for a panel of cytokines, caspases and growth factors using ELISA will be monitored.

GROUPS / COHORTS (4):
- chronic HCV: chronic HCV either treated or not with DAAs.Flow cytometry and Western Blot analysis for each subgroup
  Interventions: Diagnostic Test: Flow cytometry and Western Blot analysis
- Liver cirrhosis without HCC: Liver cirrhosis without HCC either received treatment or not.Flow cytometry and Western Blot analysis for each subgroup
  Interventions: Diagnostic Test: Flow cytometry and Western Blot analysis
- Liver cirrhosis with HCC: Liver cirrhosis with HCC either received treatment or not.Flow cytometry and Western Blot analysis for each subgroup
  Interventions: Diagnostic Test: Flow cytometry and Western Blot analysis
- Control group: Healthy subjects

INTERVENTIONS:
Diagnostic Test: Flow cytometry and Western Blot analysis — Diagnostic tests
  Groups: Liver cirrhosis with HCC; Liver cirrhosis without HCC; chronic HCV

SUMMARY:
Case control Study to assess the difference of immune cell responses between patients with chronic HCV- related liver cirrhosis who develop HCC after treatment with DAAs and those who do not develop HCC

DETAILED DESCRIPTION:
Clinical and laboratory assessment with measurement of Child-Pugh and MELD scores to assess the severity of liver disease and measurement of alpha fetoprotein level for HCC cases will be done.

Radiological assessment using abdominal ultrasound and triphasic CT will be done to determine the extent of the HCC and staging.

Blood sample from all patients will be withdrawn. Plasma will be isolated and stored at - 20C and further analysis for a panel of cytokines, caspases and growth factors using ELISA will be monitored.

Peripheral blood mononuclear cells (PBMCs) will be isolated using ficoll gradient method and will then be stored at -80C.

B and T cell proliferation in response to specific antigens will also be investigated using CFSE staining assay followed by flow cytometry analysis for CD4, CD8 and PD-1.

Cell cycle analysis and apoptosis will be detected using Annexin V/PI staining method and flow cytometry analysis. The phosphorylation and activation of cytoplasmic proteins will be tested using Western blot analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC on top of HCV related liver cirrhosis either received treatment or not
* Patients without HCC either received treatment or not .
* Patients with chronic HCV as a control group either received treatment or not.

Exclusion Criteria:

* Patients with HCC who received any interventional treatment as alcohol injection, radiofrequency , TACE..etc
* Patients with recurrent HCC after curative treatment.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cases recruited divided into three groups .Each group either treated or not with DAAs
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Pattern of immunity in patients with de novo HCC develped after treatment with DAAs | Two months
  Difference of B and T cells immune responses after treatment with DAAs between those who develop HCC and those who do not develop HCC

CONTACTS AND LOCATIONS:
Overall Officials: Haidi Ramadan, Lecturer, Principal Investigator — Lecturer
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No